CLINICAL TRIAL: NCT05316506
Title: Choose Your Words Wisely: Impact of a Provider's Language on Perceived Pain During Office Hysteroscopy: A Randomized Controlled Trial
Brief Title: Pain and Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jose Carugno, Associate Professor Obstetrics and Gynecology Minimally Invasive Gynecology/Robotic Division Director., University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20211092
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hysteroscopy Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticipated Discomfort Group (Other): Participants will be prompted using anticipated discomfort language during the standard of care hysteroscopy.
  Interventions: Other: Anticipated Discomfort Language
- Objective Description Group (Other): Participants will be prompted using objective description language during the standard of care hysteroscopy.
  Interventions: Other: Objective Descriptive Language

INTERVENTIONS:
Other: Anticipated Discomfort Language — This language involves pain descriptors provided from physician to patient during procedure.
  Arms: Anticipated Discomfort Group
Other: Objective Descriptive Language — This language involves neutral/objective descriptors provided from physician to patients during procedure.
  Arms: Objective Description Group

SUMMARY:
The purpose of this research is to look at the impact that phrases of likely discomfort or a description of the procedure have on the perception of pain during in-office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older
2. Scheduled for in office hysteroscopy
3. Able to consent for the study in English or Spanish

Exclusion Criteria:

1. Persons with preexisting conditions that may alter pain perception (ie. active vulvo-vaginal infection, vulvodynia, genital lesions, chronic pain conditions)
2. Previous in-office hysteroscopy
3. Hysteroscopy for foreign body/ Intrauterine Device (IUD) removal
4. Minors, prisoners, or other members of vulnerable populations
5. Patients who cannot communicate in English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain as measured by Visual Analog Scale (VAS) | Baseline (pre-procedure), Day 1 (post-procedure)
  Pain will be assessed using the Visual Analog Scale (VAS). Visual Analog Scale (VAS) is score from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Number of participants in each pain category | Day 1 (post-procedure)
  Number of participants reporting actual pain compared to their anticipated the pain post procedure.
  1. Pain Free
  2. Less painful than anticipated
  3. As painful as anticipated
  4. More painful than anticipated
  5. Much more painful than anticipated

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carugno, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No